CLINICAL TRIAL: NCT04449757
Title: Fluid Resuscitation Management for Patients With Septic Shock: the Efficacy and Safety Comparison Between Bicarbonated Ringer's Solution and Lactated Ringer's Solution
Brief Title: Bicarbonated Ringer's Solution Versus Lactated Ringer's Solution in Patients With Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, ZhiYong Peng, Professor; Chief physician, Zhongnan Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2020044
Record Dates: First submitted 2020-05-27; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Septic Shock; Fluid Resuscitation; Crystalloid Solution; Intensive Care Unit
Keywords: septic shock; fluid resuscitation; crystalloid solution; intensive care unit
MeSH Terms: conditions — Shock, Septic | interventions — bicarbonated Ringer's solution; Ringer's Lactate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bicarbonated ringer's solution (Experimental): We apply bicarbonated ringer's solution as resuscitation fluid to patients with septic shock.
  Interventions: Drug: Bicarbonated Ringer's solution
- lactated ringer's solution (Experimental): We apply lactated ringer's solution as resuscitation fluid to patients with septic shock.
  Interventions: Drug: Lactated Ringer's solution

INTERVENTIONS:
Drug: Bicarbonated Ringer's solution — Method of administration: intravenous infusion; 500-1000ml each time; Speed of infusion: it is decided by the clinicians.
  Other Names: Ringers Bicarbonate
  Arms: bicarbonated ringer's solution
Drug: Lactated Ringer's solution — Method of administration: intravenous infusion; 500-1000ml each time; Speed of infusion: it is decided by the clinicians.
  Other Names: Ringers Lactate
  Arms: lactated ringer's solution

SUMMARY:
In this prospective randomized controlled trial, investigators aim to study the effects and safety of bicarbonated Ringer's solution in patients with septic shock compared with lactated ringer's solution, and provide evidence for current fluid resuscitation strategies for septic shock.

DETAILED DESCRIPTION:
Although the latest guidelines recommend crystalloids as the first choice for the patients' fluid resuscitation, it still remains controversial that which crystalloid solution is the best choice. It is reported that balanced crystalloid can result in better outcomes than saline for critically ill patients. However, there are few studies conducted between different crystalloid solutions.

Lactated ringer's solution is the longest-used crystalloid solution. Compared with lactated ringer's solution whose anion is lactate, the anion of bicarbonate ringer's solution is bicarbonate. And lactate needs to be metabolized into bicarbonate through the mitochondria of the liver before it can play an alkalization role. Therefore, in theory, bicarbonate ringer's solution does not need to rely on liver metabolism, the onset time to maintain acid-base balance is shorter, and it may be more suitable for patients with severe acidosis. In patients with septic shock, the incidence of moderate to severe metabolic is increased. Bicarbonate ringer's solution can directly supplement the concentration of bicarbonate, while lactated ringer's solution needs to take time and be metabolized in the liver. Thus, we hypothesize that bicarbonate ringer's solution is more effective for patients with shock and metabolic acidosis than lactated ringer's solution.

ELIGIBILITY:
Inclusion Criteria:

* 1. At the age of 18 to 75;
* 2. Being treated in the ICU;
* 3. Diagnosed as septic shock according tho the definition of Sepsis 3.0 with fluid resuscitation requirement.

Exclusion Criteria:

* 1. Severe hepatic failure;
* 2. Possible brain injury;
* 3. With absolute contraindications for central vena catheterization;
* 4. Ever participated in another clinical trial within 30 days prior enrollment;
* 5. Have corrected metabolic acidosis through alkaline drug application within 24 hours prior to enrollment;
* 6. Hypermagnesemia or hypothyroidism;
* 7. Pregnant of breast-feeding women;
* 8. Considered inevitable death;
* 9. Other situations where investigators think enrollment is not appropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
the average doses of vasopressors | From the onset of shock to the first blood pressure stabilization (MAP≥65mmHg), or serum lactate <2.2mmol/l, or discontinuation of vasoactive drugs. About 24 hours.
  total doses of norepinephrine÷weight÷duration of usage

SECONDARY OUTCOMES:
the PH value | 0, 3 hours, 6 hours, 12 hours, 24 hours
  the potencial of hydrogen of arterial blood
the BE value | 0, 3 hours, 6 hours, 12 hours, 24 hours
  the base excess of arterial blood
shock reversal time | From the onset of shock to the first blood pressure stabilization (MAP≥65mmHg), or serum lactate <2.2mmol/l, or discontinuation of vasoactive drugs. About 24 hours.
  From the onset of shock to the first blood pressure stabilization (MAP≥65mmHg), or serum lactate <2.2mmol/l, or discontinuation of vasoactive drugs
total volume of fluids before hemodynamic stabilization | From the onset of shock to the first blood pressure stabilization (MAP≥65mmHg), or serum lactate <2.2mmol/l, or discontinuation of vasoactive drugs. About 24 hours.
  total volume of bicarbonated ringers/lactated ringers before hemodynamic stabilization
the change of serum lactate value at the 6th hour | 6 hours
  serum lactate (6h) - serum lactate (0h)
the proportion of patients whose serum lactate decreases 30% | From the onset of shock to the first blood pressure stabilization (MAP≥65mmHg), or serum lactate <2.2mmol/l, or discontinuation of vasoactive drugs. About 24 hours.
  the proportion of patients whose serum lactate decreases 30%
mortality from any cause | on the day28 after enrollment
  the rate of death from any cause within 28 days after enrollment
the rate of metabolic alkalosis | From the onset of shock to the first blood pressure stabilization (MAP≥65mmHg), or serum lactate <2.2mmol/l, or discontinuation of vasoactive drugs. About 24 hours.
  the percentage of metabolic alkalosis (PH>7.45 and HCO3>26mmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided